CLINICAL TRIAL: NCT01092169
Title: Prevalence Of Microalbuminuria Among Children Suffering From Sickle Cell Nephropathy and Sickle Cell/Beta-Thalassemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Amit Hochberg, Pediatrics Department, Hillel Yaffe Medical Center
Other Study IDs: 64/2009
Record Dates: First submitted 2010-03-23; First posted 2010-03-24 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2010-03

CONDITIONS: Sickle Cell Anemia; Beta-Thalassemia; Microalbuminuria
MeSH Terms: conditions — Anemia, Sickle Cell; beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Sickle cell beta
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Sickle cell nephropathy is a known complication of sickle cell anemia (SCA) manifested by increase in glomerular filtration rate (glomerular hyperfiltration) and results in proteinuria and chronic renal failure.

Our goal is to examine the prevalence of proteinuria and microalbuminuria as an early predictive factor of glomerular injury, among young people who suffer from SCA as well as those who suffer from combined sickle cell/beta-thalassemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sickle cell anemia
* Patients diagnosed with combined sickle cell anemia/beta-thalassemia

Exclusion Criteria:

* Diabetes mellitus
* Hypertension
* Reduced renal mass (single kidney)
* Overweight
* History of UTIs

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Young people suffering from SCA as well as those who suffer from combined sickle cell/beta-thalassemia, between 0-25 years old.
Sampling Method: Non-Probability Sample